CLINICAL TRIAL: NCT03179111
Title: Evaluation of Low Pressure Pneumoperitoneum in Bariatric Surgery: A Prospective Randomized Study
Brief Title: Evaluation of Low Pressure Pneumoperitoneum in Bariatric Surgery (ELOPES Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Tikfu Gee, Principle Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR-16-1488-32135 (IIR)
Record Dates: First submitted 2017-05-24; First posted 2017-06-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Surgical View; Shoulder Tip Pain; Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Intervention Model Description: There will be two arms in this study. One arm will be the low pressure pneumoperitoneum group (8-10mmHg) where else the other arm will be the standard pressure pneumoperitoneum group (12-15mmHg).
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study. Neither the participant (patient) nor the investigator (surgeon) will know which group the particular participant will be assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Pressure Group (Experimental): Participants will undergo elective bariatric surgery. Participants under this group will be given intra-abdominal pressure of 8-10mmHg. The number of subjects anticipated for this arm will be 47. Participants in this low pressure group are expected to encounter lesser shoulder tip pain and abdominal pain. Operating field for surgeons also expected to be better.
  Interventions: Procedure: Pneumoperitoneum Pressure
- Standard Pressure Group (Experimental): Participants will undergo elective bariatric surgery. Participants under this group will be given intra-abdominal pressure of 12-15mmHg. The number of subjects anticipated for this arm will be 47. Participants in this group are expected to have an increased amount of shoulder tip pain and higher pain score postoperatively compared to low pressure group. Operating fields for surgeons are expected to be less clear.
  Interventions: Procedure: Pneumoperitoneum Pressure

INTERVENTIONS:
Procedure: Pneumoperitoneum Pressure — There will be two arms in this study. The participants recruited for this study are those who have been screened and planned for elective bariatric surgery.The pneumoperitoneum pressure will be adjusted to either 8-10mmHg or 12-15mmHg until a clear operating field is obtained by the surgeon. Low pneumoperitoneum pressure has been expected to give a clearer and better surgical view than standard pneumoperitoneum pressure. Participants under the low pressure group are expected to have lesser pain score on abdominal pain and shoulder tip pain as compared to participants in the standard pressure group.

SUMMARY:
This is a prospective study whereby it involves patients who are planned for bariatric surgery. In the bariatric surgery procedure, pneumoperitoneum pressure will be the experimental aspect in this study. The pneumoperitoneum pressure will be adjusted to either 8-10 mmHg of low pressure or to 12-15mmHg of standard pressure.

DETAILED DESCRIPTION:
This will be a prospective study in patients aged between 18 and 70 years old who have already been screened and planned for elective bariatric surgery. In bariatric surgery, a large portion of the stomach will be removed. Pneumoperitoneum is also known as the abdominal pressure which will be the experimental aspect in this study. Laparoscopy surgery will be performed by introducing the camera (optical trocar) after making an incision at the belly button (umbilicus), and carbon dioxide which will be given at a rate of 5 L/min until the intra-abdominal pressure of either 8-10 mmHg (low-pressure group) or 12-15 mmHg (standard pressure group) is achieved. The remaining three standard ports will be placed and the laparoscopic sleeve gastrectomy will be performed at an insufflation rate of 15 L/min. The greater omentum will be divided at the greater curvature of the stomach using an ultrasonic dissector, beginning from the proximal antrum until the fundus. The omentum will be divided close to the stomach wall hence preserving the gastro-epiploic vessels. Short gastric vessels will be divided entirely from the stomach and this dissection will continue until the left crus of the diaphragm are exposed. Endoscopic staplers will then be used to staple and divide the stomach until the angle of His. A 39Fr gastric calibration tube will be placed along the lesser curvature of the stomach, acts as a guide during the division of the stomach. Finally, the divided stomach will be removed through a 12mm port site and the incision will be closed with sutures.

Towards the end of the surgery, all residual pneumoperitoneum will be evacuated by keeping the trocar valves open under direct telescopic vision. The duration of surgery or any intraoperative complications will be recorded. The starting of surgery will be regarded after the induction of anaesthesia and the end of surgery is regarded when the end of skin closure. Operating field or also known as surgical view is defined as the view of the intra-abdomen. A clear operating field allows a good working space for the surgeon. Numeric rating score will be used to access the operating field during the surgery. Post-operative pain will be rated on a Visual Analog Scale at rest and with movement.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Ability to give informed consent
* Patients who are approved by the anaesthetics to undergo bariatric surgery.

Exclusion Criteria:

* Age below 18 and above 70
* Inability to give informed consent
* Patient unfit for bariatric surgery including who has poor respiratory, cardiac, renal and liver function.
* Patient with Body Mass Index (BMI) >50
* Patient with American Society of Anesthesiologists (ASA) >3

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Operating Field | It will be assessed intraoperatively (during the surgery).
  Numeric rating score will be used to access the operating field during the surgery. The numeric rating score will be recorded after the surgery by the surgeon. The score ranges from 1 to 4 whereby 1 means poor space with excessive muscular contractions and unable to proceed with surgery safely. Numeric rating scale of 4 indicates good surgical space. If there was any compromise of the operating field (NOS score ≥ 3), the pneumoperitoneum pressure will be increased accordingly.

SECONDARY OUTCOMES:
Pain Score | The abdomen and shoulder tip pain intensity will be rated up to 48 hours postoperatively.
  The pain score will be assessed using visual analog scale (VAS) (0-10). A score of 0 means no pain, whereas a score of 10 equals the worst pain ever experienced. Post-operative pain will be rated on a visual analog score at rest. The time of arrival in the postoperative recovery room will be defined as zero hours postoperatively. The patients will be asked about the location of pain, whether at the shoulder, incision sites, and/or inside the abdomen by the medical doctors or nurses.
Duration of Surgery | The starting of surgery will be regarded after the induction of anaesthesia and the end of surgery is regarded when the end of skin closure.
  The duration of surgery or any intraoperative complications will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Lindekaer AL, Riber C, Gatke MR. Surgical space conditions during low-pressure laparoscopic cholecystectomy with deep versus moderate neuromuscular blockade: a randomized clinical study. Anesth Analg. 2014 Nov;119(5):1084-92. doi: 10.1213/ANE.0000000000000316. PMID 24977638
- [Background] Neudecker J, Sauerland S, Neugebauer E, Bergamaschi R, Bonjer HJ, Cuschieri A, Fuchs KH, Jacobi Ch, Jansen FW, Koivusalo AM, Lacy A, McMahon MJ, Millat B, Schwenk W. The European Association for Endoscopic Surgery clinical practice guideline on the pneumoperitoneum for laparoscopic surgery. Surg Endosc. 2002 Jul;16(7):1121-43. doi: 10.1007/s00464-001-9166-7. Epub 2001 May 20. PMID 12015619
- [Background] Litynski GS. Kurt Semm and an automatic insufflator. JSLS. 1998 Apr-Jun;2(2):197-200. PMID 9876740
- [Background] Ibraheim OA, Samarkandi AH, Alshehry H, Faden A, Farouk EO. Lactate and acid base changes during laparoscopic cholecystectomy. Middle East J Anaesthesiol. 2006 Feb;18(4):757-68. PMID 16749570
- [Background] Schietroma M, Carlei F, Mownah A, Franchi L, Mazzotta C, Sozio A, Amicucci G. Changes in the blood coagulation, fibrinolysis, and cytokine profile during laparoscopic and open cholecystectomy. Surg Endosc. 2004 Jul;18(7):1090-6. doi: 10.1007/s00464-003-8819-0. Epub 2004 May 12. PMID 15136925
- [Background] Esmat ME, Elsebae MM, Nasr MM, Elsebaie SB. Combined low pressure pneumoperitoneum and intraperitoneal infusion of normal saline for reducing shoulder tip pain following laparoscopic cholecystectomy. World J Surg. 2006 Nov;30(11):1969-73. doi: 10.1007/s00268-005-0752-z. PMID 17043939
- [Background] Schietroma M, Pessia B, Stifini D, Lancione L, Carlei F, Cecilia EM, Amicucci G. Effects of low and standard intra-abdominal pressure on systemic inflammation and immune response in laparoscopic adrenalectomy: A prospective randomised study. J Minim Access Surg. 2016 Apr-Jun;12(2):109-17. doi: 10.4103/0972-9941.178513. PMID 27073301
- [Background] Gurusamy KS, Vaughan J, Davidson BR. Low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 18;2014(3):CD006930. doi: 10.1002/14651858.CD006930.pub3. PMID 24639018
- [Background] Nguyen NT, Wolfe BM. The physiologic effects of pneumoperitoneum in the morbidly obese. Ann Surg. 2005 Feb;241(2):219-26. doi: 10.1097/01.sla.0000151791.93571.70. PMID 15650630
- [Background] Buunen M, Gholghesaei M, Veldkamp R, Meijer DW, Bonjer HJ, Bouvy ND. Stress response to laparoscopic surgery: a review. Surg Endosc. 2004 Jul;18(7):1022-8. doi: 10.1007/s00464-003-9169-7. Epub 2004 May 12. PMID 15136930
- [Background] Gupta A, Watson DI. Effect of laparoscopy on immune function. Br J Surg. 2001 Oct;88(10):1296-306. doi: 10.1046/j.0007-1323.2001.01860.x. PMID 11578282
- [Background] Sylla P, Kirman I, Whelan RL. Immunological advantages of advanced laparoscopy. Surg Clin North Am. 2005 Feb;85(1):1-18, vii. doi: 10.1016/j.suc.2004.09.005. PMID 15619524
- [Background] Hajri A, Mutter D, Wack S, Bastien C, Gury JF, Marescaux J, Aprahamian M. Dual effect of laparoscopy on cell-mediated immunity. Eur Surg Res. 2000;32(5):261-6. doi: 10.1159/000008773. PMID 11111169
- [Background] West MA, Baker J, Bellingham J. Kinetics of decreased LPS-stimulated cytokine release by macrophages exposed to CO2. J Surg Res. 1996 Jun;63(1):269-74. doi: 10.1006/jsre.1996.0259. PMID 8661209
- [Background] Umar A, Mehta KS, Mehta N. Evaluation of hemodynamic changes using different intra-abdominal pressures for laparoscopic cholecystectomy. Indian J Surg. 2013 Aug;75(4):284-9. doi: 10.1007/s12262-012-0484-x. Epub 2012 May 1. PMID 24426454
- [Background] Kelman GR, Swapp GH, Smith I, Benzie RJ, Gordon NL. Caridac output and arterial blood-gas tension during laparoscopy. Br J Anaesth. 1972 Nov;44(11):1155-62. doi: 10.1093/bja/44.11.1155. No abstract available. PMID 4265051
- [Background] Helmy SA, Wahby MA, El-Nawaway M. The effect of anaesthesia and surgery on plasma cytokine production. Anaesthesia. 1999 Aug;54(8):733-8. doi: 10.1046/j.1365-2044.1999.00947.x. PMID 10460524
- [Background] Carlei F, Schietroma M, Cianca G, Risetti A, Mattucci S, Ngome Enang G, Simi M. Effects of laparoscopic and conventional (open) cholecystectomy on human leukocyte antigen-DR expression in peripheral blood monocytes: correlations with immunologic status. World J Surg. 1999 Jan;23(1):18-22. doi: 10.1007/s002689900559. PMID 9841758
- [Background] Schietroma M, Carlei F, Cappelli S, Amicucci G. Intestinal permeability and systemic endotoxemia after laparotomic or laparoscopic cholecystectomy. Ann Surg. 2006 Mar;243(3):359-63. doi: 10.1097/01.sla.0000201455.89037.f6. PMID 16495701
- [Background] Schietroma M, Carlei F, Rossi M, Mattucci S, Gulla N, Lezoche E. Neutrophil-elastase in patients undergoing open versus laparoscopic cholecystectomy. Surgery. 2001 Nov;130(5):898. doi: 10.1067/msy.2001.117374. No abstract available. PMID 11685204
- [Background] Visser BC, Parks RW, Garden OJ. Open cholecystectomy in the laparoendoscopic era. Am J Surg. 2008 Jan;195(1):108-14. doi: 10.1016/j.amjsurg.2007.04.008. PMID 18082551
- [Background] Torres K, Torres A, Staskiewicz GJ, Chroscicki A, Los T, Maciejewski R. A comparative study of angiogenic and cytokine responses after laparoscopic cholecystectomy performed with standard- and low-pressure pneumoperitoneum. Surg Endosc. 2009 Sep;23(9):2117-23. doi: 10.1007/s00464-008-0234-0. Epub 2008 Dec 6. PMID 19067057
- [Background] Basgul E, Bahadir B, Celiker V, Karagoz AH, Hamaloglu E, Aypar U. Effects of low and high intra-abdominal pressure on immune response in laparoscopic cholecystectomy. Saudi Med J. 2004 Dec;25(12):1888-91. PMID 15711660
- [Background] Ozdemir-van Brunschot DM, van Laarhoven KC, Scheffer GJ, Pouwels S, Wever KE, Warle MC. What is the evidence for the use of low-pressure pneumoperitoneum? A systematic review. Surg Endosc. 2016 May;30(5):2049-65. doi: 10.1007/s00464-015-4454-9. Epub 2015 Aug 15. PMID 26275545
- [Background] Mann C, Boccara G, Pouzeratte Y, Eliet J, Serradel-Le Gal C, Vergnes C, Bichet DG, Guillon G, Fabre JM, Colson P. The relationship among carbon dioxide pneumoperitoneum, vasopressin release, and hemodynamic changes. Anesth Analg. 1999 Aug;89(2):278-83. doi: 10.1097/00000539-199908000-00003. PMID 10439730
- [Background] Arnolda L, McGrath BP, Johnston CI. Vasopressin and angiotensin II contribute equally to the increased afterload in rabbits with heart failure. Cardiovasc Res. 1991 Jan;25(1):68-72. doi: 10.1093/cvr/25.1.68. PMID 2054832
- [Background] Feig BW, Berger DH, Dougherty TB, Dupuis JF, Hsi B, Hickey RC, Ota DM. Pharmacologic intervention can reestablish baseline hemodynamic parameters during laparoscopy. Surgery. 1994 Oct;116(4):733-9; discussion 739-41. PMID 7940173
- [Background] Hypolito OH, Azevedo JL, de Lima Alvarenga Caldeira FM, de Azevedo OC, Miyahira SA, Miguel GP, Becker OM Jr, Machado AC, Nunes Filho GP, Azevedo GC. Creation of pneumoperitoneum: noninvasive monitoring of clinical effects of elevated intraperitoneal pressure for the insertion of the first trocar. Surg Endosc. 2010 Jul;24(7):1663-9. doi: 10.1007/s00464-009-0827-2. Epub 2009 Dec 25. PMID 20035347
- [Background] Vijayaraghavan N, Sistla SC, Kundra P, Ananthanarayan PH, Karthikeyan VS, Ali SM, Sasi SP, Vikram K. Comparison of standard-pressure and low-pressure pneumoperitoneum in laparoscopic cholecystectomy: a double blinded randomized controlled study. Surg Laparosc Endosc Percutan Tech. 2014 Apr;24(2):127-33. doi: 10.1097/SLE.0b013e3182937980. PMID 24686347
- [Background] Obeid F, Saba A, Fath J, Guslits B, Chung R, Sorensen V, Buck J, Horst M. Increases in intra-abdominal pressure affect pulmonary compliance. Arch Surg. 1995 May;130(5):544-7; discussion 547-8. doi: 10.1001/archsurg.1995.01430050094016. PMID 7748095
- [Background] O'Leary E, Hubbard K, Tormey W, Cunningham AJ. Laparoscopic cholecystectomy: haemodynamic and neuroendocrine responses after pneumoperitoneum and changes in position. Br J Anaesth. 1996 May;76(5):640-4. doi: 10.1093/bja/76.5.640. PMID 8688262
- [Background] Davides D, Birbas K, Vezakis A, McMahon MJ. Routine low-pressure pneumoperitoneum during laparoscopic cholecystectomy. Surg Endosc. 1999 Sep;13(9):887-9. doi: 10.1007/s004649901126. PMID 10449845
- [Background] Rosin D, Brasesco O, Varela J, Saber AA, You S, Rosenthal RJ, Cohn SM. Low-pressure laparoscopy may ameliorate intracranial hypertension and renal hypoperfusion. J Laparoendosc Adv Surg Tech A. 2002 Feb;12(1):15-9. doi: 10.1089/109264202753486876. PMID 11905857
- [Background] Wallace DH, Serpell MG, Baxter JN, O'Dwyer PJ. Randomized trial of different insufflation pressures for laparoscopic cholecystectomy. Br J Surg. 1997 Apr;84(4):455-8. PMID 9112891
- [Background] Kim MH, Lee KY, Lee KY, Min BS, Yoo YC. Maintaining Optimal Surgical Conditions With Low Insufflation Pressures is Possible With Deep Neuromuscular Blockade During Laparoscopic Colorectal Surgery: A Prospective, Randomized, Double-Blind, Parallel-Group Clinical Trial. Medicine (Baltimore). 2016 Mar;95(9):e2920. doi: 10.1097/MD.0000000000002920. PMID 26945393
- [Background] Blobner M, Frick CG, Stauble RB, Feussner H, Schaller SJ, Unterbuchner C, Lingg C, Geisler M, Fink H. Neuromuscular blockade improves surgical conditions (NISCO). Surg Endosc. 2015 Mar;29(3):627-36. doi: 10.1007/s00464-014-3711-7. Epub 2014 Aug 15. PMID 25125097
- [Background] Barczynski M, Herman RM. A prospective randomized trial on comparison of low-pressure (LP) and standard-pressure (SP) pneumoperitoneum for laparoscopic cholecystectomy. Surg Endosc. 2003 Apr;17(4):533-8. doi: 10.1007/s00464-002-9121-2. Epub 2003 Feb 17. PMID 12582754